CLINICAL TRIAL: NCT00884429
Title: Effectiveness of Chest Physiotherapy Actual Versus Conventional Techniques in Infants With Acute Viral Bronchiolitis. Random Clinical Trial
Brief Title: Effectiveness of Chest Physiotherapy in Infants With Acute Viral Bronchiolitis
Acronym: ECPAVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Evelim Leal de Freitas Dantas Gomes, Master in Science Rehabilitation, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHSL
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-01

CONDITIONS: Viral Bronchiolitis
Keywords: Chest physiotherapy
MeSH Terms: conditions — Bronchiolitis, Viral

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1- Conventional Chest Physiotherapy (Active Comparator): Percussion , thorax compression and Postural Drainage/suction if necessary
  Interventions: Procedure: Chest physiotherapy - Conventional
- 2- Chest physiotherapy- Actual techniques (Active Comparator): slow prolonged expiration and clearance rhinopharynx and suction if necessary
  Interventions: Procedure: Chest physiotherapy - actual techniques
- 3- Airway Suction (Active Comparator): Suction superior airways. Only in admission.
  Interventions: Procedure: 3-Airway suction

INTERVENTIONS:
Procedure: Chest physiotherapy - Conventional — Percussion Postural Drainage and thorax compression
  Arms: 1- Conventional Chest Physiotherapy
Procedure: Chest physiotherapy - actual techniques — Slow prolonged expiration and clearance rhinopharynx retrograde
  Arms: 2- Chest physiotherapy- Actual techniques
Procedure: 3-Airway suction — Airway suction
  Arms: 3- Airway Suction

SUMMARY:
The purpose of this study is to verify the effectiveness of chest physiotherapy (actual versus conventional) on respiratory distress in infants with acute viral bronchiolitis.

DETAILED DESCRIPTION:
The infants were random in three groups: Conventional techniques, actual techniques and suction of upper airways On the first two groups the infants were evaluated on admission,48,72hours and before hospital discharge. On third group was evaluated only on admission when SRV was collected.

Respiratory distress was evaluated with Wang's score by the physiotherapists and nurses not participating in the research.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute viral bronchiolitis
* RSV positive

Exclusion Criteria:

* Heart diseases
* Chronic lung disease
* Neurological diseases
* Parental refusal
* Previous wheezing episode
* ventilatory support

Ages: 28 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Respiratory distress | on first evaluation by physiotherapyst ( until 2 hours after hospital admission)
  This outcome was evaluated with Wang's score for infants with bronchiolitis

SECONDARY OUTCOMES:
Respiratory distress | 48 hours after first evaluation
  Wang's score
Respiratory distress | 72 hours after first evaluation
  Wang's score
Respiratory distress | 1 hour before hospital discharge
  wang's score

CONTACTS AND LOCATIONS:
Overall Officials: Evelim LF Dantas Gomes, Master, Principal Investigator — Hospital Sírio Libanês e UNINOVE
Locations (1):
- Hospital Sírio Libanês, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196
- [Derived] Gomes EL, Postiaux G, Medeiros DR, Monteiro KK, Sampaio LM, Costa D. Chest physical therapy is effective in reducing the clinical score in bronchiolitis: randomized controlled trial. Rev Bras Fisioter. 2012 Jun;16(3):241-7. doi: 10.1590/s1413-35552012005000018. Epub 2012 Apr 12. PMID 22499404